CLINICAL TRIAL: NCT07213375
Title: High Dose Dexamethasone In High-Pain Responders Undergoing Enhanced Recovery Video-Assisted Thoracoscopic Surgery Lobectomy and Segmentectomy - A Randomized Double-Blinded Controlled Trial
Brief Title: High Dose Dexamethasone to Reduce Postoperative Pain After Video-Assisted Thoracoscopic Surgery Lobectomy /Segmentectomy
Acronym: DEXTER
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lasse Visby, Co-investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-520891-25-00; 2025-520891-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Analgetic; Lung Cancer (NSCLC); Video Assisted Thoracic Surgery (VATS); Glucocorticoid
Keywords: Pain catastrophizing; ERAS; VATS; Lung cancer; Minimizing pain
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose Dexamethasone (8mg) (Active Comparator)
  Interventions: Drug: Dexamethasone
- High dose Dexamethasone (1mg/kg) (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Patients will receive either low dose (8mg) or high dose (1mg/kg)

SUMMARY:
The aim is to conduct a randomized controlled trial (RCT) with a high dose arm (1mg/kg) vs a low dose (8mg in total) of steroid (Dexamethasone) given intravenous (IV) after the induction of anesthesia to "High-pain-responders" in patients undergoing VATS lobectomy/segmentectomy.

The hypothesis is that a high dose of Dexamethasone can lower pain when coughing in the morning after VATS lobectomy/segmentectomy, in patients scoring as "High-pain-responders" on the Pain-Catastrophizing-Scale

DETAILED DESCRIPTION:
Annually, approximately 400 anatomical resections (lobectomy and segmentectomy) are performed using video-assisted thoracoscopic surgery (VATS) at the Department of Cardiothoracic Surgery, Rigshospitalet.

Tissue damage occurs during surgery, triggering an inflammatory response.Glucocorticoids, including Dexamethasone, administered in relation to surgery, have shown anti-inflammatory effects in previous studies and the potential to reduce postoperative pain and hospitalization duration in various surgical procedures.

Previous studies have indicated that the most common complications of VATS lobectomy leading to prolonged hospitalization in patients are air leakage (27%), pneumonia (20%), and pain (15%).

A previous study from Rigshospitalet, Denmark found that half of the patients undergoing a VATS lobectomy, reported severe pain (defined as Numeric Rating Scale (NRS) ≥ 5) at some point on the day of surgery and first postoperative day. This indicates a need for better pain management following VATS lobectomy, which is confirmed by another study Rigshospitalet, Denmark that found a high rate of severe pain (NRS > 5) in the first two days after a VATS lobectomy. The median NRS score when coughing on the morning after surgery was 6.0 (5.0-8.0). Improved pain management is expected to facilitate easier mobilization, likely resulting in fewer pulmonary complications and shorter hospital stays.

The Pain Catastrophizing Scale (PCS) is a self-assessment questionnaire examining catastrophic thinking in relation to pain. The PCS score has previously been shown to correlate with postoperative pain, and in another study found that increasing scores of PCS resulted in higher pain scores, and that patients grouped as "High-pain-responders" (PCS≥20) had significantly more pain when coughing on the first postoperative day.

Previous studies, in patients undergoing a total knee arthroplasty, showed that higher doses of Dexamethasone reduced the percentage of patients experiencing moderate-severe pain postoperatively in the "High-pain-responder" group, however not in the "Low-pain-responder" group.

The aim is to conduct a randomized controlled trial (RCT) with a high dose arm (1mg/kg) vs a low dose (8mg in total) of steroid (Dexamethasone) given intravenous (IV) after the induction of anesthesia to "High-pain-responders" in patients undergoing VATS lobecto-my/segmentectomy.

Safety of higher doses of glucocorticoid has previously been extensively examined and side effects are considered negligible, and several larger meta-analyses of previous studies have only minor side effects with glucocorticoids in both low and high doses when compared to placebo.

Previous studies have also performed exactly the same intervention, with same doses of Dexamethasone, in patients scheduled for knee and hip arthroplasty without any safety issues.

The hypothesis is that a high dose of Dexamethasone can lower pain when coughing in th morning after VATS lobectomy/segmentectomy, in patients scoring as "High-pain-responders" on the Pain-Catastrophizing-Scale

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Able to understand written and spoken Danish language
* PCS ≥20
* Signed written informed consent form.
* Patient planned to elective VATS lobectomy/segmentectomy

Exclusion Criteria:

* Patients undergoing systemic glucocorticoid or other immunosuppressive therapies, ex-cluding inhaled steroids.

  * Individuals with diabetes requiring insulin treatment.
  * Pregnant or breastfeeding patients.
  * Patients with known allergies to the study drug.
  * Individuals with mental disabilities that may impair their capacity to provide informed consent or compromise the validity of data collection.
  * Patients with diagnosed schizophrenia, active psychosis, bipolar disorder, or a history of ongoing treatment with antipsychotic and/or antidepressant medications.
  * Individuals with altered pain perception due to other conditions or injuries, such as spi-nal cord or brain injuries, severe polyneuropathies, or neurological disorders.
  * Regular users of opioid medications.
  * Patients requiring reoperation within the first two postoperative days.
  * Individuals undergoing conversion to a surgical procedure other than VATS lobecto-my/segmentectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain when coughing on the morning of first postoperative day. | Morning of first postoperative day
  The primary endpoint is pain when coughing on the first morning after surgery, measured on the NRS-scale (0-10; where 0 is no pain, and 10 is the worst possible pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Cardiothoracic Surgery, Rigshospitalet, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided